CLINICAL TRIAL: NCT02963857
Title: Evaluation of a Breast Biblock Analgesia for the Mastectomy With Radical Axillary Lymphadenectomy Surgery
Status: Completed | Type: Observational
Sponsor: Maison de Santé Prostestante de Bordeaux Bagatelle (Other)
Responsible Party: Principal Investigator, Dr Claude-Charles Balick-Weber, Claude-Charles Balick-Weber, MD, Maison de Santé Prostestante de Bordeaux Bagatelle
Other Study IDs: Evaluation of a breast biblock
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Mastectomy, Segmental; Acute Pain; Anesthesia
Keywords: breast surgery; acute pain; regional anesthesia
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the efficacy of the the pecto-intercostal fascial plane block (PIF block) for the anesthesia of the intercostal nerves anterior branches and assesses the association of the serratus block with a PIF block for the breast surgery.

DETAILED DESCRIPTION:
Breast surgery is one of the most painful post-operative surgery. This surgery is well known to induce postoperative chronic pain. The paravertebral block, because of its efficacy and less invasive nature than epidural analgesia, is quickly becoming the reference technique for pain management of major breast surgery.

Peripheral regional anesthesia for the breast surgery appeared in the past few years. Among these techniques are the PEC block, Serratus block and more recently the pecto-intercostal fascial plane block (PIF block).

Currently in the investigators hospital in every day's practice, an association of the serratus block and the PIF block is made, which allows for a complete block of both the laterals branches of intercostal nerves (with the serratus block) and of anterior branches of intercostal nerves (with the PIF block). Therefore, this association of blocks may lead to a complete analgesia of the breast, while the serratus block alone only allows for analgesia of the lateral part of the breast.

This technique was previously described. The authors evoked the possibility of the association of serratus and PIF blocks and described this technique with a patient, but to the investigators knowledge no evaluation of the efficacy of this procedure was made.

The objective of the study is to analyze this technique through a collection form that evaluates the satisfaction and post-operative morphine consumption of women receiving this association of blocks before a general anesthesia for a unilateral mastectomy with homolateral total lymphadenectomy.

This is a purely observational study that assesses a current practice in this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* total mastectomy surgery with a complete axillary lymph nodes removal

Exclusion Criteria:

* age under 18
* contraindication to the surgery
* refusal of the protocol by the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients included in the study have had a total mastectomy surgery with a complete axillary lymph nodes removal.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary goal of the study is to evaluate the postoperative morphine consumption until 72 hours after the surgery. | 3 days

SECONDARY OUTCOMES:
Pain levels on a numeric pain rating scale were recorded at rest and with arm mobilization during the first 72 hours. | 3 days
level of comfort during the first 72 hours was recorded (the 4 levels-scale used was: excellent, good, medium and bad). | 3 days

IPD SHARING:
Plan to Share IPD: No